CLINICAL TRIAL: NCT06761833
Title: The Effect of Preoperative Anxiety on Postoperative Behavioral Changes in Children Receiving Dental Treatment Under General Anesthesia
Brief Title: Postoperative Behavioral Changes in Children.
Status: Not yet recruiting | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Other Study IDs: BaskentU-EKILINC-001
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Behavior Problems; Pediatrics; Pediatric Pain and Anxiety
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single center observational study

SUMMARY:
In children scheduled for dental treatment, negative thoughts can lead to anxiety and make them resistant to treatment techniques. In our prospective, single-center observational study, we aim to investigate preoperative anxiety and postoperative negative behaviors in children aged 3 to 12 years who are set to undergo general anesthesia for dental conditions and treatments.

DETAILED DESCRIPTION:
The study will involve children aged 3 to 12 who have been classified under the American Society of Anesthesiologists (ASA) as I-II. These children, scheduled for dental treatment between January 2025 and January 2026 at Başkent University Adana's Turgut Noyan Practice and Research Hospital, will undergo elective surgery under general anesthesia. Parental consent will be obtained prior to their inclusion in the research.

The assessment of preoperative anxiety levels in patients will be conducted using the Modified Yale Preoperative Anxiety Scale (m-YPAS). This evaluation will take place in the presence of their families within the anesthesia outpatient clinic and the preoperative preparation room on the day of surgery. The m-YPAS is structured into five categories: Activity, Speech, Emotional State, Awaking State, and Parent-Related Reactions, comprising a total of 22 items. The scoring for the Modified Yale Preoperative Anxiety Scale ranges from 5 to 22 points, with each item assigned a single point. Research has demonstrated that the Turkish validation of the m-YPAS is a valid and reliable tool for assessing preoperative anxiety in children aged 5 to 12 years.

Induction of general anesthesia will be standardized for all patients. The Bispectral Index (BIS) will be kept between 40- 60. All patients will receive standard local anesthetic by the pedodontist during the operation. The anesthesia physician will evaluate delirium using the Pediatric Postoperative Delirium Scale (PAED) at 1 minute post-surgery and every 10 minutes thereafter until the patient is transferred to the ward. The PAED scale has been used in Turkish studies to assess postoperative delirium. İn the absence of complications during the patient's follow-up in the ward, the patient will be discharged on the same day. To evaluate behavioral changes in children during the preoperative period, parents will be provided with information regarding the 11 item Post-Hospital Discharge Behavior Questionnaire ( PHBQ-AS) in the outpatient clinic. Parents will be requested to compare their children's behavior prior to hospitalization with their behavior following discharge for each item on the questionnaire. Additionally, follow-up phone calls will be conducted on the 2nd, 15th, and 30th days after discharge to collect and record survey results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients categorized as American Society of Anesthesiologists (ASA) groups 1 and 2.
2. Children aged 3 to 12 years who are scheduled to receive dental treatment under general anesthesia.

Exclusion Criteria:

1. The child patient or parent has a diagnosed psychiatric disorder.
2. There is a history of substance use that may affect cognitive function.
3. The parent has declined to participate in the study.
4. The child patient or parent does not speak Turkish.
5. Patients categorized as American Society of Anesthesiologists (ASA) group 3 and 4.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients between the ages of 3 and 12 who are scheduled to receive dental treatment under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The effect of preoperative anxiety level on postoperative behavioral changes in children receiving dental treatment under general anesthesia. | one year
  This observational study, conducted at a single center, aims to investigate the occurrence of negative postoperative behavior in children

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent Universty Adana Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided